CLINICAL TRIAL: NCT00891007
Title: Partially Randomized, Controlled Phase II Study to Evaluate Safety, Dose Response and Immunogenicity of the Measles Vaccine MVA mBN85B in Healthy Children Aged 6 Months to 6 Years
Brief Title: Study to Evaluate Safety, Dose Response and Immunogenicity of the Measles Vaccine MVA mBN85B in Healthy Children Aged 6 Months to 6 Years
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bavarian Nordic (Industry)
Responsible Party: Monika Fluer, Bavarian Nordic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MEA-HFN-002
Record Dates: First submitted 2009-04-29; First posted 2009-04-30 (Estimated); Last update posted 2012-07-27 (Estimated); Status verified 2012-07

CONDITIONS: Measles
Keywords: Measles; Virus Disease; Paediatric Diseases; Paramyoxyviridae
MeSH Terms: conditions — Measles; Virus Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Experimental)
  Interventions: Biological: MVA-mBN85B
- Group 2 (Experimental)
  Interventions: Biological: MVA-mBN85B
- Group 3 (Active Comparator)
  Interventions: Biological: Rouvax

INTERVENTIONS:
Biological: MVA-mBN85B — Low Dose arm, 1x 10E7 TCID50
  Arms: Group 1
Biological: MVA-mBN85B — Normal Dose arm, 1x 10E8 TCID50
  Arms: Group 2
Biological: Rouvax — Standard measles vaccine, approved in South Africa
  Arms: Group 3

SUMMARY:
Partially randomized, controlled Phase II study to evaluate safety, immunogenicity and dose response of the measles vaccine MVA mBN85B in healthy children aged 6 months to 6 years.

DETAILED DESCRIPTION:
Open label study to assess the safety and immunogenicity of MVA-mBN85B in healthy vaccine-naive, measles-naive and measles-experienced children. The study is comprised of three groups with 30 children each. Two groups will receive two subcutaneous (s.c.) immunizations 4 weeks (28±3 days) apart of either either 1 x 10E7 TCID50 (Group A) or 1 x 10E8 TCID50 (Group B) MVA mBN85B. The control group (Group C) will receive two s.c. doses (0.5 ml, 1000 TCID50) of Rouvax® (Sanofi-Pasteur) 24 weeks apart.

ELIGIBILITY:
Inclusion Criteria:

1. Read, signed and dated informed consent document from one parent/guardian of the child after being advised of the risks and benefits of the study in a language understood by the parent/guardian. This document must be signed prior to performance of any study specific procedure.
2. Male or female child between the age of 6 months to 6 years (Group C: 9 months to 6 years).
3. Prior or no prior measles vaccination indicated on the RTHC.
4. No known exposure to measles within 30 days prior to study entry.
5. No history of measles disease.
6. Negative human immunodeficiency virus antibody test (anti-HIV) and hepatitis B surface antigen (HBsAG).
7. Child is in good health as determined by medical history, physical examination and clinical judgment.
8. Children for whom the investigator reasonably believes its parents/guardian can and will comply with the requirements of the protocol

Exclusion Criteria:

1. Any clinically significant condition that may influence participation in this study, including febrile convulsions.
2. Severe malnutrition as assessed by the investigator by weight for age and clinical criteria.
3. History of splenectomy.
4. Clinically significant anaemia (laboratory and clinical criteria).
5. Having received any vaccinations or planned vaccinations with a live vaccine within 30 days prior to or after study vaccination.
6. Having received any vaccinations or planned vaccinations with a killed vaccine within 14 days prior to or after study vaccination.
7. Administration or planned administration of immunoglobulins and/or any blood products during a period starting from 3 months prior to administration of the vaccine and ending at study conclusion.
8. Use of any investigational or non-registered drug or vaccine other than the study vaccine within 30 days preceding the first dose of the study vaccine, or planned administration of such a drug during the study period.
9. History of any serious medical condition, which in the opinion of the investigator, would compromise the safety of the child.
10. History of or currently active autoimmune disease. Children with vitiligo or thyroid disease on thyroid replacement therapy are not excluded.
11. History of malignancy, especially leukaemia or lymphoma.
12. History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
13. History of anaphylaxis or severe allergic reaction.
14. Known allergy to egg proteins, gelatine, neomycin or gentamycin.
15. Chronic administration (defined as more than 14 days) of systemic high dose immuno-suppressant drugs during a period starting from six months prior to administration of the vaccine and ending at study conclusion. High dose is defined as 2 mg/kg/day or more of prednisolone or its equivalent, or 20 mg/day or more for children who weigh more than 10 kg.
16. Previous participation in an MVA-based vaccination study

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2009-06; Primary Completion 2010-07 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Chris Hani Baragwanath Hospital, Respiratory and Meningeal Pathogens Research Unit, Bertsham, South Africa